CLINICAL TRIAL: NCT03224026
Title: Which Virus Leads to Viremia in Children With Fever Without Source and do New Biomarkers Correlate With Viral and Bacterial Infections?
Brief Title: Validation of a Proteomic Signature and Assessment of Viremia in Children With Fever Without Source
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: MM-15082-Vir
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Infectious Disease; Fever; Viremia
MeSH Terms: conditions — Communicable Diseases; Fever; Viremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fever Without Source: Clinical diagnosis of FWS (fever of less than 7 days with no cause determined by the history and the physical exam).
- Healthy control: Children visiting the hospital due to a non-infectious, non inflammatory etiology

SUMMARY:
The study is an observational blinded Validation study in pediatric patients below 3 years old with a diagnosis of Fever Without Source (FWS). In this study the investigators aim to validate the performance of a proteomic signature aiding the physicians to discriminate between viral and bacterial infections in febrile children. The study will also assess the prevalence of Human Enteroviruses (HEV), Human Parechoviruses (HPeV), Adenovirus (AdV) and Human Herpesvirus type 6 (HHV-6) viremia, as well as Kingella Kingae bacteremia in the study cohort.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of FWS (fever of less than 7 days with no cause determined by the history or the physical exam)
* Age < 3 years old
* Informed consent (IC) given by parent or legal guardian

Exclusion Criteria:

* Unavailable blood
* Comorbidities predisposing to infections such as cancer, primary or secondary immunodeficiency, and iatrogenic immunosuppression

Inclusion Criteria for healthy controls:

* Age < 3 years old
* Informed consent (IC) given by parent or legal guardian
* No suspicion of infectious or inflammatory disease at presentation and during the two weeks before.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients below three years old which were presented with a diagnosis of fever without source to the emergency room in the Children's Hospital, Geneva University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy compared to expert panel for bacterial versus viral. | 0-7 days after initiation of symptoms
  Sensitivity, specificity, NPV and PPV were measured for ImmunoXpert and Labscore.
  The proteomic signature is a combination of different markers including: tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) (pg/mL), interferon γ-induced protein-10 (IP-10) (pg/mL) and C-reactive protein (CRP) (mg/L). The proteomic signature is expressed as a score (no units. ranges 0-100).
  The Labscore is a combination of procalcitonin (ng/mL), C-reactive protein (CRP) (mg/L) and urinary dipstix (positive if presence of leucocyturia or nitrites). The Lab-score is expressed as a score (no units. ranges 0-9)

SECONDARY OUTCOMES:
Diagnostic accuracy compared to microbiology gold standard for ruling out invasive bacterial infection. | 0-7 days after initiation of symptoms
  Case by case comparison between microbiology gold standard and ImmunoXpert and Labscore.
  The proteomic signature is a combination of different markers including: tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) (pg/mL), interferon γ-induced protein-10 (IP-10) (pg/mL) and C-reactive protein (CRP) (mg/L). The proteomic signature is expressed as a score (no units, ranges 0-100).
  The Labscore is a combination of procalcitonin (ng/mL), C-reactive protein (CRP) (mg/L) and urinary dipstix (positive if presence of leucocyturia or nitrites). The Lab-score is expressed as a score (no units, ranges 0-9).
Comparison of biomarker levels in patients with different etiologies as classified by the expert panel or healthy. | 0-7 days after initiation of symptoms in cases with infection.
  An expert panel classified a patient as experiencing a bacterial versus viral infection. In addition healthy patients were requited.
  The following biomarkers were examined across the healthy versus bacterial versus viral patients:
  1. The proteomic signature is a combination of different markers including: tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) (pg/mL), interferon γ-induced protein-10 (IP-10) (pg/mL) and C-reactive protein (CRP) (mg/L). The proteomic signature is expressed as a score (no units, ranges 0-100).
  2. The Labscore is a combination of procalcitonin (ng/mL), C-reactive protein (CRP) (mg/L) and urinary dipstix (positive if presence of leucocyturia or nitrites). The Lab-score is expressed as a score (no units, ranges 0-9).
  3. Tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) (pg/mL).
  4. interferon γ-induced protein-10 (IP-10) (pg/mL).
  5. C-reactive protein (CRP) (mg/L).
Prevalence of viruses in children with fever without source. | 0-7 days after the initiation of symptoms
  Prevalence of Human Enteroviruses, Human Parechoviruses, Adenovirus and Human Herpesvirus type 6 viremia and viremia from other microorganism identified by Next-Generation Sequencing (NGS) (no units) or other techniques, as well as K. kingae bacteremia in children under three years old presenting with fever without source.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oved K, Cohen A, Boico O, Navon R, Friedman T, Etshtein L, Kriger O, Bamberger E, Fonar Y, Yacobov R, Wolchinsky R, Denkberg G, Dotan Y, Hochberg A, Reiter Y, Grupper M, Srugo I, Feigin P, Gorfine M, Chistyakov I, Dagan R, Klein A, Potasman I, Eden E. A novel host-proteome signature for distinguishing between acute bacterial and viral infections. PLoS One. 2015 Mar 18;10(3):e0120012. doi: 10.1371/journal.pone.0120012. eCollection 2015. PMID 25785720
- [Background] Colvin JM, Muenzer JT, Jaffe DM, Smason A, Deych E, Shannon WD, Arens MQ, Buller RS, Lee WM, Weinstock EJ, Weinstock GM, Storch GA. Detection of viruses in young children with fever without an apparent source. Pediatrics. 2012 Dec;130(6):e1455-62. doi: 10.1542/peds.2012-1391. Epub 2012 Nov 5. PMID 23129086
- [Background] Ambrosioni J, Bridevaux PO, Wagner G, Mamin A, Kaiser L. Epidemiology of viral respiratory infections in a tertiary care centre in the era of molecular diagnosis, Geneva, Switzerland, 2011-2012. Clin Microbiol Infect. 2014 Sep;20(9):O578-84. doi: 10.1111/1469-0691.12525. Epub 2014 Jan 24. PMID 24382326
- [Derived] L'Huillier AG, Mardegan C, Cordey S, Luterbacher F, Papis S, Hugon F, Kaiser L, Gervaix A, Posfay-Barbe K, Galetto-Lacour A. Enterovirus, parechovirus, adenovirus and herpes virus type 6 viraemia in fever without source. Arch Dis Child. 2020 Feb;105(2):180-186. doi: 10.1136/archdischild-2019-317382. Epub 2019 Aug 28. PMID 31462437